CLINICAL TRIAL: NCT00524407
Title: The Effects of PROCRIT (Epoetin Alfa) on Hemoglobin, Symptom Distress, and Quality of Life During Chemotherapy in Lymphoma, Chronic Lymphocytic Leukemia or Multiple Myeloma Patients With Mild to Moderate Anemia
Brief Title: Effect of Epoetin Alfa on Hemoglobin, Symptom Distress, and Quality of Life in Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho Biotech, Inc. (Industry)
Organization: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005125
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Chemotherapy; Anemia; Cancer
Keywords: Anemia; hemoglobin; chemotherapy; hematologic response; subcutaneous injection; Epoetin alfa; FACT-An; LASA; PROCRIT
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study was to compare the effectiveness of epoetin alfa treatment on hemoglobin (Hb) response, quality of life (QoL), health care resource utilization and patient productivity when epoetin alfa was administered during chemotherapy to patients with mild anemia or after waiting until patients became moderately anemic. Patients with lymphoma, chronic lymphocytic leukemia (CLL) or Multiple Myeloma (MM) were studied.

DETAILED DESCRIPTION:
This study was an open-label (patients and investigators knew what treatment was being given), randomized (patients were assigned to a treatment group by chance) study of lymphoma, chronic lymphocytic leukemia (CLL), or multiple myeloma patients. This study addressed the clinical and patient-management consequences of treating mild to moderate anemia (hemoglobin (Hb) between 10 and 12 g/dL). The design of the study compared the effect of treating higher Hb levels to current standard of care criteria on Hb levels, transfusion requirements, and patient reported outcomes (quality of life, health care resource utilization, and productivity). Patients were randomized according to their Hb levels. Two entry criteria were specified during the course of the trial. Initially, patients were enrolled with Hb levels >= 11 g/dL and then randomized to receive 1) Immediate epoetin alfa treatment or 2) Observed after Hb levels fell below 11 g/dL. Epoetin alfa treatment was provided to the Observed group if and when Hb levels fell below 9.0 g/dL. Slow recruitment of patients in to the study resulted in a protocol amendment. Subsequently, if a patient presented with a Hb between 10 and 12 g/dL, the patient was randomized to the Immediate or to the Observed groups. Patients presenting with Hgb > 12 g/dL but otherwise eligible, were not randomized until Hb dropped to <=12 g/dL. Patients remained in the study for up to 36 weeks. Safety assessments were performed throughout the study and included obtaining and evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events. The starting dose of PROCRIT (Epoetin alfa) was administered subcutaneously (sc) as 40,000 Units (U) once weekly (qw). If after 3-4 weeks of therapy, the Hb did not increase by > 1.0 g/dL, the dose was increased to 60,000 U sc qw. If at any time, the Hb rose above 15 g/dL on 2 consecutive evaluations, PROCRIT (Epoetin alfa) was stopped until the Hb dropped to below 13 g/dL and then resumed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must present with non-Hodgkins Lymphoma (Low, Intermediate or High Grade) or Hodgkins Disease, CLL or Multiple Myeloma
* Life expectancy > 6 months with Karnofsky Performance Index of > =70
* Evaluable lesion as objective indicator of response
* Scheduled for at least one myelosuppressive cytotoxic regimen (experimental chemotherapy allowed) for at least 4-6 months
* Patients with reproductive potential must have used an adequate contraceptive method
* Transferrin saturation = 20% and serum ferritin = 50 ng/mL Bone marrow evaluations may be performed to determine if iron stores are adequate
* histologic documentation of disease.

Exclusion Criteria:

* Patients with no second active malignancy or history of other malignancy diagnosed within preceding 5 years (other than basal cell carcinoma or cervical cancer)
* No uncontrolled hypertension
* active, unresolved infection
* anemia due to factors other than cancer/chemotherapy, i.e., iron, folate, hemolysis, or GI bleeding
* Receiving Epoetin alfa independent of protocol
* Received chemotherapy with the previous 14 days
* Prior total lymphoid, extensive abdominal or inverted Y radiation therapy
* No use of interferons or interleukins during study
* No use of nonchemotherapy experimental agents within preceding 30 days
* No Hodgkins Disease patients who are chemotherapy naïve
* Received stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 1996-07; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
To measure the change in quality of life score as demonstrated by the FACT-An (Functional Assessment in Cancer Therapy - Anemia) and LASA (Linear Analogue Assessment Scale) tools over the 36 week study period.

SECONDARY OUTCOMES:
Health care resource utilization. To measure transfusion requirements and change in Hb levels. All patients were followed for survival until closure of study which was the time the last patient in the entire study completed study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech, Inc. Clinical Trial, Study Director — Ortho Biotech, Inc.

REFERENCES:
- [Result] Straus DJ, Testa MA, Sarokhan BJ, Czuczman MS, Tulpule A, Turner RR, Riggs SA. Quality-of-life and health benefits of early treatment of mild anemia: a randomized trial of epoetin alfa in patients receiving chemotherapy for hematologic malignancies. Cancer. 2006 Oct 15;107(8):1909-17. doi: 10.1002/cncr.22221. PMID 16977654